CLINICAL TRIAL: NCT06655818
Title: A Phase I/II, Randomized, Open-label Platform Study Utilizing a Master Protocol to Study Belantamab Mafodotin (GSK2857916) as Monotherapy and in Combination With Anti-Cancer Treatments in Participants With Relapsed/Refractory Multiple Myeloma (RRMM)-DREAMM5. Sub-study 4 - Belantamab Mafodotin and Dostarlimab (GSK4057190) in Combination
Brief Title: Sub-study of Belantamab Mafodotin (GSK2857916) as Monotherapy and in Combination With Dostarlimab (GSK4057190) in Participants With RRMM
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to lack of efficacy
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 208887 Sub Study 4; 2019-001138-32 (EudraCT Number)
Expanded Access: NCT03763370 (Available)
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Results first posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Relapsed/Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — belantamab mafodotin; dostarlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Belantamab mafodotin + Dostarlimab (Experimental)
  Interventions: Drug: Belantamab Mafodotin; Drug: Dostarlimab

INTERVENTIONS:
Drug: Belantamab Mafodotin — Belantamab Mafodotin will be administered.
  Other Names: GSK2857916
Drug: Dostarlimab — Dostarlimab will be administered.
  Other Names: GSK4057190

SUMMARY:
The primary purpose is to determine the safety and tolerability of belantamab mafodotin in combination with other anti-cancer treatments (in each sub-study), and to establish the recommended Phase 2 dose for each combination treatment to explore in the cohort expansion phase. This study is a sub study of the Master protocol (NCT04126200).

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 years of age inclusive or older, at the time of signing the informed consent.
* Participants must have histologically or cytologically confirmed diagnosis of Multiple Myeloma (MM), as defined by the IMWG.
* Participants having at least 3 prior lines of prior anti-myeloma treatments including an immunomodulating agent (IMID) a proteasome inhibitor (PI) and an anti-CD38 monoclonal antibody.
* Participants with a history of autologous stem cell transplant are eligible for study participation when, transplant was >100 days prior to study enrolment and with no active infection(s).
* Participants with Eastern Cooperative Oncology Group (ECOG) performance status of 0-1, unless ECOG less than equal to (<=)2 is due solely to skeletal complications and/or skeletal pain due to MM.
* Participants with measurable disease defined as at least one of the following: Serum M-protein greater than equal to (>=)0.5 gram per deciliter (>=5 gram per liter) or Urine M-protein >=200 milligrams (mg) per 24 hours or Serum free light chain (FLC) assay: Involved FLC level >=10 mg per deciliter (>=100 mg per Liter) and an abnormal serum FLC ratio (<0.26 or >1.65).
* Participants who have tested positive for Hepatitis B core antibody (HBcAb) can be enrolled if the following criteria are met: Serology result HBcAb+, Hepatitis B surface antigen (HBsAg)-; HBV deoxyribonucleic acid (DNA) undetectable during screening.
* Participants who are currently receiving physiological doses oral steroids (<10 mg/day), inhaled steroids or ophthalmological steroids.

Exclusion Criteria:

* Participants with current corneal epithelial disease except mild punctate keratopathy.
* Participants with evidence of cardiovascular risk.
* Participants with known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to belantamab mafodotin or any of the components of the study treatment. History of severe hypersensitivity to other mAb.
* Participants with active infection requiring antibiotic, antiviral, or antifungal treatment.
* Participants with other monoclonal antibodies within 30 days or systemic anti-myeloma therapy within <14 days.
* Participants with prior radiotherapy within 2 weeks of start of study therapy.
* Participants with prior allogeneic transplant are prohibited.
* Participants who have received prior Chimeric Antigen T cell therapy (CAR-T) therapy with lymphodepletion with chemotherapy within 3 months of screening.
* Participants with any major surgery (other than bone-stabilizing surgery) within the last 30 days.
* Participants with prior treatment with an investigational agent within 14 days or 5 half-lives of receiving the first dose of study drugs, whichever is shorter.
* Participants with >=grade 3 toxicity considered related to prior check-point inhibitors and that led to treatment discontinuation.
* Participants who have received transfusion of blood products within 2 weeks before the first dose of study drug.
* Participants must not receive live attenuated vaccines within 30 days prior to first dose of study treatment or whilst receiving belantamab mafodotin +- partner agent in any sub-study arm of the platform trial and for at least 70 days following last study treatment.
* Participants with presence of active renal condition (infection, requirement for dialysis or any other condition that could affect participant's safety). Participants with isolated proteinuria resulting from MM.
* Participants with known human immunodeficiency virus (HIV) infection, unless the participant can meet all criteria: a) established anti-retroviral therapy for at least 4 weeks and HIV viral load<400 copies/milliliter (mL) b) cluster of differentiation 4 plus (CD4+) T-cell (CD4+) counts >= 350 cells/microliter (µL) c) No history of Acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections within the last 12 months in which case the participant would be eligible for CE Phase only.
* Participants with autoimmune disease (current or history) or syndrome that required systemic treatment within the past 2 years.
* Exclusion for a recent (within the past 6 months) history of symptomatic pericarditis.
* Participant has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs).
* Participants who have received prior therapy with an anti-programmed death-1 (anti-PD-1), anti-PD-1-ligand-1 (anti-PD-L1), or anti-PD-1 ligand-2 (anti-PD-L2) agent.
* Participant has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment. Use of inhaled steroids, local injection of steroids, and steroid eye drops are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- GSK Investigational Site, Lille, France
- South Korea (2):
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Ulsan

IPD SHARING:
Plan to Share IPD: No
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a sub study of the master study NCT04126200. This sub study was terminated due to lack of efficacy. The study was planned to include two phases - Dose Escalation (DE) and Cohort Expansion (CE) and no participants from this sub study were enrolled in CE phase as study was early terminated.
Groups:
- 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab: Participants with Relapsed/Refractory Multiple Myeloma (RRMM) received 1.9 milligram (mg)/kilogram (kg) belantamab mafodotin intravenous (IV) infusion as powder for solution once every 3 weeks (Q3W) infused over 30- 60 minutes on day 1 of 21-day cycles in combination with 500 mg dostarlimab as a 30-minute IV infusion 1 hour after belantamab mafodotin end of infusion (EOI) on day 1 of 21-day cycles (Q3W).
Period: Overall Study
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Started | 4
Completed (Participants who completed follow-up or who died were considered to have completed the study.) | 3 (1 participant completed the follow-up and 2 participants died.)
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: YEAR] | 70.0 (9.83)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Gender categories (with 0<n<11) are combined into 'Males and Females' category to maintain participant confidentiality and privacy as the study is evaluating a rare disease.
  Participants
    Males and Females | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race categories (with 0<n<11) are combined into 'Others' category to maintain participant confidentiality and privacy as the study is evaluating a rare disease.
  Participants
    Others | 4

OUTCOME MEASURES:

1. Primary Outcome: DE Phase: Number of Participants With Dose Limiting Toxicities (DLT)
Description: Criteria for dose-limiting toxicity (DLT) included hematologic indicators such as Grade 3-5 febrile neutropenia and thrombocytopenia with bleeding. Non-hematologic criteria, excluding corneal toxicity, comprise Grade 3-5 toxicities, with exceptions for manageable nausea, vomiting, or diarrhea, controlled Grade 3 hypertension, and events linked to disease progression. Tumor lysis syndrome (TLS) of Grade 3 or 4, successfully managed within 7 days without end-organ damage, is considered. Corneal toxicity, assessed by the GSK corneal grading scale at Grade 4, is a DLT. Other organ-specific toxicities, notably liver toxicity meeting GSK stopping criteria, also qualify as DLTs. Severity was graded using National Cancer Institute - Common Terminology Criteria for Adverse Events (version 5.0).
Time Frame: Up to 21 days
Population: DLT Evaluable Population included participants in DE who have received the first course of treatment containing both agents within a sub-study and followed up within cycle 1 (Each cycle is of 21 days) or withdrew within cycle 1 due to an AE meeting the definition of a DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 4
Participants | 1

2. Primary Outcome: DE Phase: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AEs were coded using the Medical Dictionary for Regulatory Activities (MedDRA) coding system.
Time Frame: Up to 153 weeks
Population: Safety population included all participants who received at least 1 dose of any component of the combination therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 4
Participants | 4

3. Primary Outcome: DE Phase: Number of Participants With Worst-Case Hematology Results by Maximum Grade Increase Post - Baseline Relative to Baseline
Description: Blood samples were collected for the analysis of following hematology parameters: eosinophils, anemia, hemoglobin increased, lymphocyte count decreased, lymphocyte count increased, neutrophil count decreased, platelet count decreased, leukocytosis and white blood cell decreased. Grade 1 (G1): mild; Grade 2 (G2): moderate; Grade 3 (G3): severe; Grade 4 (G4) life-threatening or disabling. Higher grade indicates greater severity and an increase in CTCAE grade was defined relative to the Baseline grade. Any worst-case post baseline increase to G1, G2, G3, and G4 are presented. The laboratory parameters were graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.
Time Frame: Baseline (Day 1) and up to 153 weeks
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 4
Participants
  Eosinophilia, Increase to Grade 1 | 0
  Eosinophilia, Increase to Grade 2 | 0
  Eosinophilia, Increase to Grade 3 | 0
  Eosinophilia, Increase to Grade 4 | 0
  Anemia, Increase to Grade 1 | 0
  Anemia, Increase to Grade 2 | 1
  Anemia, Increase to Grade 3 | 1
  Anemia, Increase to Grade 4 | 0
  Hemoglobin increased, Increase to Grade 1 | 0
  Hemoglobin increased, Increase to Grade 2 | 1
  Hemoglobin increased, Increase to Grade 3 | 0
  Hemoglobin increased, Increase to Grade 4 | 0
  Lymphocyte count decreased, Increase to Grade 1 | 0
  Lymphocyte count decreased, Increase to Grade 2 | 0
  Lymphocyte count decreased, Increase to Grade 3 | 0
  Lymphocyte count decreased, Increase to Grade 4 | 2
  Lymphocyte count increased, Increase to Grade 1 | 0
  Lymphocyte count increased, Increase to Grade 2 | 1
  Lymphocyte count increased, Increase to Grade 3 | 0
  Lymphocyte count increased, Increase to Grade 4 | 0
  Neutrophil count decreased, Increase to Grade 1 | 0
  Neutrophil count decreased, Increase to Grade 2 | 1
  Neutrophil count decreased, Increase to Grade 3 | 1
  Neutrophil count decreased, Increase to Grade 4 | 1
  Platelet count decreased, Increase to Grade 1 | 1
  Platelet count decreased, Increase to Grade 2 | 0
  Platelet count decreased, Increase to Grade 3 | 2
  Platelet count decreased, Increase to Grade 4 | 0
  Leukocytosis, Increase to Grade 1 | 0
  Leukocytosis, Increase to Grade 2 | 0
  Leukocytosis, Increase to Grade 3 | 0
  Leukocytosis, Increase to Grade 4 | 0
  White blood cell decreased, Increase to Grade 1 | 0
  White blood cell decreased, Increase to Grade 2 | 0
  White blood cell decreased, Increase to Grade 3 | 0
  White blood cell decreased, Increase to Grade 4 | 1

4. Primary Outcome: DE Phase: Number of Participants With Worst-Case Chemistry Results by Maximum Grade Increase Post - Baseline Relative to Baseline
Description: Blood samples were collected for the analysis of following chemistry parameters: Hypoglycemia, hypoalbuminemia, alkaline phosphatase (ALP) increased, alanine aminotransferase (ALT) increased, aspartate aminotransferase (AST) increased, blood bilirubin increased, creatine kinase (CPK) increased, creatinine increased, gamma glutamyl transferase (GGT) increased, hyperkalemia, blood lactate dehydrogenase (LDH) increased, hypermagnesemia, hypomagnesemia, hypernatremia, hypercalcemia, hypocalcemia and chronic kidney disease. G1: mild; G2: moderate; G3: severe. Higher grade indicates greater severity and an increase in CTCAE grade was defined relative to the Baseline grade. Any worst-case post baseline increase to G1, G2 and G3 are presented. The laboratory parameters were graded according to CTCAE version 5.
Time Frame: Baseline (Day 1) and up to 153 weeks
Population: Safety Population. Only those participants with data available at the specified categories were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 4
Participants
  Hypoglycemia, Increase to Grade 1 | 0
  Hypoglycemia, Increase to Grade 2 | 0
  Hypoglycemia, Increase to Grade 3 | 0
  Hypoalbuminemia, Increase to Grade 1 | 0
  Hypoalbuminemia, Increase to Grade 2 | 2
  Hypoalbuminemia, Increase to Grade 3 | 0
  Alkaline phosphatase increased, Increase to Grade 1 | 0
  Alkaline phosphatase increased, Increase to Grade 2 | 0
  Alkaline phosphatase increased, Increase to Grade 3 | 0
  Alanine aminotransferase increased, Increase to Grade 1 | 2
  Alanine aminotransferase increased, Increase to Grade 2 | 1
  Alanine aminotransferase increased, Increase to Grade 3 | 0
  Aspartate aminotransferase increased, Increase to Grade 1 | 2
  Aspartate aminotransferase increased, Increase to Grade 2 | 0
  Aspartate aminotransferase increased, Increase to Grade 3 | 1
  Blood bilirubin increased, Increase to Grade 1 | 0
  Blood bilirubin increased, Increase to Grade 2 | 1
  Blood bilirubin increased, Increase to Grade 3 | 0
  CPK increased, Increase to Grade 1: number analyzed (Participants) | 3
  CPK increased, Increase to Grade 1 | 1
  CPK increased, Increase to Grade 2: number analyzed (Participants) | 3
  CPK increased, Increase to Grade 2 | 0
  CPK increased, Increase to Grade 3: number analyzed (Participants) | 3
  CPK increased, Increase to Grade 3 | 0
  Creatinine increased, Increase to Grade 1 | 2
  Creatinine increased, Increase to Grade 2 | 0
  Creatinine increased, Increase to Grade 3 | 0
  GGT increased, Increase to Grade 1 | 1
  GGT increased, Increase to Grade 2 | 0
  GGT increased, Increase to Grade 3 | 0
  Hyperkalemia, Increase to Grade 1 | 0
  Hyperkalemia, Increase to Grade 2 | 0
  Hyperkalemia, Increase to Grade 3 | 0
  Blood lactate dehydrogenase increased, Increase to Grade 1 | 4
  Blood lactate dehydrogenase increased, Increase to Grade 2 | 0
  Blood lactate dehydrogenase increased, Increase to Grade 3 | 0
  Hypermagnesemia, Increase to Grade 1: number analyzed (Participants) | 3
  Hypermagnesemia, Increase to Grade 1 | 1
  Hypermagnesemia, Increase to Grade 2: number analyzed (Participants) | 3
  Hypermagnesemia, Increase to Grade 2 | 0
  Hypermagnesemia, Increase to Grade 3: number analyzed (Participants) | 3
  Hypermagnesemia, Increase to Grade 3 | 0
  Hypomagnesemia, Increase to Grade 1: number analyzed (Participants) | 3
  Hypomagnesemia, Increase to Grade 1 | 0
  Hypomagnesemia, Increase to Grade 2: number analyzed (Participants) | 3
  Hypomagnesemia, Increase to Grade 2 | 0
  Hypomagnesemia, Increase to Grade 3: number analyzed (Participants) | 3
  Hypomagnesemia, Increase to Grade 3 | 0
  Hypernatremia, Increase to Grade 1 | 0
  Hypernatremia, Increase to Grade 2 | 0
  Hypernatremia, Increase to Grade 3 | 0
  Hypercalcemia, Increase to Grade 1 | 1
  Hypercalcemia, Increase to Grade 2 | 0
  Hypercalcemia, Increase to Grade 3 | 0
  Hypocalcemia, Increase to Grade 1 | 0
  Hypocalcemia, Increase to Grade 2 | 0
  Hypocalcemia, Increase to Grade 3 | 0
  Chronic Kidney Disease, Increase to Grade 1: number analyzed (Participants) | 2
  Chronic Kidney Disease, Increase to Grade 1 | 0
  Chronic Kidney Disease, Increase to Grade 2: number analyzed (Participants) | 2
  Chronic Kidney Disease, Increase to Grade 2 | 0
  Chronic Kidney Disease, Increase to Grade 3: number analyzed (Participants) | 2
  Chronic Kidney Disease, Increase to Grade 3 | 0

5. Primary Outcome: CE Phase: Overall Response Rate (ORR)
Description: Overall Response Rate (ORR) was defined as the percentage of participants with a confirmed PR or better as the best overall response (i.e., Partial Response [PR], Very Good Partial Response [VGPR], Complete Response [CR], and stringent Complete Response [sCR]), as assessed by the investigator per international myeloma working group (IMWG) (2016). CR defined as negative immunofixation of serum and urine AND disappearance of any soft tissue plasmacytomas AND <5% plasmacytomas in the bone marrow; sCR defined as CR as above PLUS normal serum free light-chain (FLC) assay ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence; VGPR defined as serum and urine M-component detectable by immunofixation but not on electrophoresis OR ≥ 90% reduction in serum M-component plus urine M-component <100 mg/24 h; PR defined as ≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥90% or to <200 mg/24 h.
Time Frame: Up to 26 weeks
Population: No participants were enrolled in CE Phase as study was terminated.
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 0

6. Secondary Outcome: DE Phase: Overall Response Rate (ORR)
Description: as for outcome 5
Time Frame: Up to 153 weeks
Population: Safety Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 4
Percentage of participants | 25 [0.6 to 80.6]

7. Secondary Outcome: CE Phase: Clinical Benefit Rate (CBR)
Description: Clinical benefit rate was defined as the percentage of participants with a confirmed minimal response (MR) or better according to the IMWG Response Criteria. MR is >= 25% but < 49% reduction of serum M-protein and reduction in 24-hour urinary M-protein by 50-89%.
Time Frame: Up to 153 weeks
Population: No participants were enrolled in CE Phase as study was terminated.
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 0

8. Secondary Outcome: DE Phase: Percentage of Participants Achieving Stringent Complete Response (SCR), Complete Response (CR), Very Good Partial Response (VGPR) and Partial Response (PR)
Description: Partial Response [PR], Very Good Partial Response [VGPR], Complete Response [CR], and stringent Complete Response [sCR] as assessed by the investigator per IMWG (2016). CR defined as negative immunofixation of serum and urine AND disappearance of any soft tissue plasmacytomas AND <5% plasmacytomas in the bone marrow; sCR defined as CR as above PLUS normal serum free light-chain (FLC) assay ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence; VGPR defined as serum and urine M-component detectable by immunofixation but not on electrophoresis OR ≥ 90% reduction in serum M-component plus urine M-component <100 mg/24 h; PR defined as ≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥90% or to <200 mg/24 h.
Time Frame: Up to 153 weeks
Population: Safety Population
Measure: Number; unit: Percentage of participants
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 4
Percentage of participants
  Stringent Complete Response (sCR) | 0
  Complete Response (CR) | 0
  Very Good Partial Response (VGPR) | 25
  Partial Response (PR) | 0

9. Secondary Outcome: CE Phase: Percentage of Participants Achieving SCR, CR, VGPR and PR
Description: Partial Response [PR], Very Good Partial Response [VGPR], Complete Response [CR], and stringent Complete Response [sCR] as assessed by the investigator per IMWG (2016). CR = negative immunofixation of serum and urine AND disappearance of any soft tissue plasmacytomas AND <5% plasmacytomas in the bone marrow; sCR=stringent complete response, CR as above PLUS normal serum free light-chain (FLC) assay ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence; VGPR = serum and urine M-component detectable by immunofixation but not on electrophoresis OR ≥ 90% reduction in serum M-component plus urine M-component <100 mg/24 h; PR = ≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥90% or to <200 mg/24 h.
Time Frame: Up to 153 weeks
Population: No participants were enrolled in CE Phase as study was terminated.
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 0

10. Secondary Outcome: DE Phase: Belantamab Mafodotin Concentrations for Plasma Antibody-Drug Conjugate (ADC)
Description: Blood samples were collected for PK analysis of belantamab mafodotin Antibody-Drug Conjugate (ADC) when administered intravenously in combination with dostarlimab.
Time Frame: Predose, end of infusion (EOI), 2, and 24 hours postdose on Cycle 1 Day 1, and at Cycle 1 Day 4, Day 8, Day 22, Predose and EOI on Cycle 2 Day 1, Cycle 4 Day 1, and at end of treatment (approximately 153 weeks)
Population: Pharmacokinetic population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Nanogram/ millilitre (ng/mL)
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 4
Nanogram/ millilitre (ng/mL)
  CYCLE 1 DAY 1, PRE-DOSE | 0.0 [0 to 0]
  CYCLE 1 DAY 1, END OF INFUSION | 25300.0 [15800 to 32300]
  CYCLE 1 DAY 1, 2 HOURS | 26450.0 [17900 to 31100]
  CYCLE 1 DAY 1, 24 HOURS | 20400.0 [8030 to 22200]
  CYCLE 1 DAY 4 | 9110.0 [5100 to 14500]
  CYCLE 1 DAY 8 | 4830.0 [2040 to 6990]
  CYCLE 1 DAY 22: number analyzed (Participants) | 1
  CYCLE 1 DAY 22 | 0.0
  CYCLE 2 DAY 1, PRE-DOSE: number analyzed (Participants) | 2
  CYCLE 2 DAY 1, PRE-DOSE | 1295.0 [1050 to 1540]
  CYCLE 2 DAY 1, END OF INFUSION: number analyzed (Participants) | 2
  CYCLE 2 DAY 1, END OF INFUSION | 41950.0 [35000 to 48900]
  CYCLE 4 DAY 1, PRE-DOSE: number analyzed (Participants) | 1
  CYCLE 4 DAY 1, PRE-DOSE | 0.0
  CYCLE 4 DAY 1, END OF INFUSION: number analyzed (Participants) | 1
  CYCLE 4 DAY 1, END OF INFUSION | 27600.0
  END OF TREATMENT: number analyzed (Participants) | 1
  END OF TREATMENT | 0.0

11. Secondary Outcome: DE Phase: Belantamab Mafodotin Concentrations for Plasma Total Antibody
Description: Blood samples were collected for PK analysis of belantamab mafodotin total antibody when administered intravenously in combination with dostarlimab.
Time Frame: as for outcome 10
Population: Pharmacokinetic population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 4
ng/mL
  CYCLE 1 DAY 1, PRE-DOSE: number analyzed (Participants) | 3
  CYCLE 1 DAY 1, PRE-DOSE | 0.0 [0 to 0]
  CYCLE 1 DAY 1, END OF INFUSION | 31000.0 [20700 to 34500]
  CYCLE 1 DAY 1, 2 HOURS | 32400.0 [19800 to 41100]
  CYCLE 1 DAY 1, 24 HOURS: number analyzed (Participants) | 3
  CYCLE 1 DAY 1, 24 HOURS | 21400.0 [12600 to 23600]
  CYCLE 1 DAY 4 | 15000.0 [7810 to 17800]
  CYCLE 1 DAY 8 | 8235.0 [4530 to 12000]
  CYCLE 1 DAY 22: number analyzed (Participants) | 1
  CYCLE 1 DAY 22 | 1140.0
  CYCLE 2 DAY 1, PRE-DOSE: number analyzed (Participants) | 2
  CYCLE 2 DAY 1, PRE-DOSE | 3625.0 [3480 to 3770]
  CYCLE 2 DAY 1, END OF INFUSION: number analyzed (Participants) | 2
  CYCLE 2 DAY 1, END OF INFUSION | 45350.0 [35500 to 55200]
  CYCLE 4 DAY 1, PRE-DOSE: number analyzed (Participants) | 1
  CYCLE 4 DAY 1, PRE-DOSE | 2800.0
  CYCLE 4 DAY 1, END OF INFUSION: number analyzed (Participants) | 1
  CYCLE 4 DAY 1, END OF INFUSION | 48900.0
  END OF TREATMENT: number analyzed (Participants) | 1
  END OF TREATMENT | 628.0

12. Secondary Outcome: DE Phase: Belantamab Mafodotin Concentrations for Plasma Cys-mcMMAF
Description: Blood samples were collected for PK analysis of belantamab mafodotin cys-mcMMAF when administered intravenously in combination with dostarlimab.
Time Frame: as for outcome 10
Population: Pharmacokinetic population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 4
ng/mL
  CYCLE 1 DAY 1, PRE-DOSE | 0.00 [0.0 to 0.0]
  CYCLE 1 DAY 1, END OF INFUSION | 218.00 [147.0 to 447.0]
  CYCLE 1 DAY 1, 2 HOURS | 376.00 [231.0 to 556.0]
  CYCLE 1 DAY 1, 24 HOURS | 750.00 [547.0 to 1670.0]
  CYCLE 1 DAY 4 | 549.50 [218.0 to 1780.0]
  CYCLE 1 DAY 8 | 170.90 [67.1 to 264.0]
  CYCLE 1 DAY 22: number analyzed (Participants) | 1
  CYCLE 1 DAY 22 | 0.00
  CYCLE 2 DAY 1, PRE-DOSE: number analyzed (Participants) | 2
  CYCLE 2 DAY 1, PRE-DOSE | 0.00 [0.0 to 0.0]
  CYCLE 2 DAY 1, END OF INFUSION: number analyzed (Participants) | 2
  CYCLE 2 DAY 1, END OF INFUSION | 555.00 [394.0 to 716.0]
  CYCLE 4 DAY 1, PRE-DOSE: number analyzed (Participants) | 1
  CYCLE 4 DAY 1, PRE-DOSE | 0.00
  CYCLE 4 DAY 1, END OF INFUSION: number analyzed (Participants) | 1
  CYCLE 4 DAY 1, END OF INFUSION | 469.00
  END OF TREATMENT: number analyzed (Participants) | 1
  END OF TREATMENT | 0.00

13. Secondary Outcome: CE Phase: Plasma Concentrations of Belantamab Mafodotin Antibody-Drug Conjugate (ADC)
Description: Blood samples were to be collected for PK analysis of Belantamab Mafodotin Antibody-Drug Conjugate (ADC).
Time Frame: Up to 153 weeks
Population: No participants were enrolled in CE Phase as study was terminated.
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 0

14. Secondary Outcome: CE Phase: Plasma Concentration of Belantamab Mafodotin Plasma Total Antibody
Description: Blood samples were to be collected for PK analysis of Belantamab mafodotin plasma total antibody.
Time Frame: Up to 153 weeks
Population: No participants were enrolled in CE Phase as study was terminated.
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 0

15. Secondary Outcome: CE Phase: Plasma Concentrations of Belantamab Mafodotin Cys- Monomethyl Auristatin-F (Cys-mcMMAF)
Description: Blood samples were to be collected for PK analysis of Belantamab Mafodotin Cys- Monomethyl Auristatin-F (Cys-mcMMAF)
Time Frame: Up to 153 weeks
Population: No participants were enrolled in CE Phase as study was terminated.
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 0

16. Secondary Outcome: DE Phase: Dostarlimab Concentration When Administered in Combination With Belantamab Mafodotin
Description: Blood samples were collected for PK analysis of dostarlimab when administered intravenously in combination with belantamab mafodotin.
Time Frame: Predose and end of infusion (EOI) on Cycle 1 Day 1, Cycle 2 Day 1, Cycle 5 Day 1, and at the end of treatment (approximately 153 weeks)
Population: Pharmacokinetic population included all participants in the Safety population who had at least 1 non-missing PK assessment. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 4
ng/mL
  CYCLE 1 DAY 1, PRE-DOSE | 0.0 [0 to 203000]
  CYCLE 1 DAY 1, END OF INFUSION | 52500.0 [0 to 124000]
  CYCLE 2 DAY 1, PRE-DOSE: number analyzed (Participants) | 2
  CYCLE 2 DAY 1, PRE-DOSE | 43550.0 [23900 to 63200]
  CYCLE 2 DAY 1, END OF INFUSION: number analyzed (Participants) | 2
  CYCLE 2 DAY 1, END OF INFUSION | 224000.0 [149000 to 299000]
  CYCLE 5 DAY 1, PRE-DOSE: number analyzed (Participants) | 1
  CYCLE 5 DAY 1, PRE-DOSE | 532.0
  CYCLE 5 DAY 1, END OF INFUSION: number analyzed (Participants) | 1
  CYCLE 5 DAY 1, END OF INFUSION | 312000.0
  END OF TREATMENT: number analyzed (Participants) | 2
  END OF TREATMENT | 35750.0 [12200 to 59300]

17. Secondary Outcome: CE Phase: Dostarlimab Concentration When Administered in Combination With Belantamab Mafodotin
Description: Blood samples were to be collected for PK analysis of dostarlimab when administered intravenously in combination with belantamab mafodotin.
Time Frame: Up to 153 weeks
Population: No participants were enrolled in CE Phase as study was terminated.
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 0

18. Secondary Outcome: DE Phase: Number of Participants With Post-baseline Positive Anti-drug Antibodies (ADAs) Against Belantamab Mafodotin
Description: Serum samples were collected for the analysis of the presence of ADAs using validated immunoassays. All samples were tested in screening assay, and positive samples were further characterized for antibody titers.
Time Frame: Up to 153 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 4
Participants | 1

19. Secondary Outcome: CE Phase: Number of Participants With Post-baseline Positive ADAs Against Belantamab Mafodotin
Description: Serum samples were to be collected for the analysis of the presence of ADAs using validated immunoassays. All samples were to be further tested in screening assay, and positive samples were further to be characterized for antibody titers.
Time Frame: Up to 153 weeks
Population: No participants were enrolled in CE Phase as study was terminated.
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 0

20. Secondary Outcome: DE Phase: Number of Participants With Post-baseline Positive ADAs Against Dostarlimab
Description: as for outcome 18
Time Frame: Up to 153 weeks
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 4
Participants | 0

21. Secondary Outcome: CE Phase: Number of Participants With Post-baseline Positive ADAs Against Dostarlimab
Description: as for outcome 19
Time Frame: Up to 153 weeks
Population: No participants were enrolled in CE Phase as study was terminated.
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 0

22. Secondary Outcome: DE Phase: Concentration of ADAs Against Dostarlimab When Administered in Combination With Belantamab Mafodotin
Description: Serum samples were collected for the analysis of the presence of ADAs using validated immunoassays. All samples were to be further tested in screening assay, and positive samples were further to be characterized for antibody titers.
Time Frame: Up to 153 weeks
Population: Safety Population. No participants were found positive for ADAs, hence participants were not analyzed for concentration of ADAs.
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 0

23. Secondary Outcome: CE Phase: Concentration of ADAs Against Dostarlimab When Administered in Combination With Belantamab Mafodotin
Description: as for outcome 19
Time Frame: Up to 153 weeks
Population: No participants were enrolled in CE Phase as study was terminated.
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 0

24. Secondary Outcome: DE Phase: Concentration of ADAs Against Belantamab Mafodotin
Description: as for outcome 22
Time Frame: Up to 153 weeks
Population: Safety Population. Only those participants with positive post-baseline antibody against belantamab mafodotin were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 1
ng/mL | NA (NA) — Data was not estimable for 1 participant as the values were below the level of detection

25. Secondary Outcome: CE Phase: Concentration of ADAs Against Belantamab Mafodotin
Description: as for outcome 19
Time Frame: Up to 153 weeks
Population: No participants were enrolled in CE Phase as study was terminated.
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 0

26. Secondary Outcome: DE Phase: Number of Participants With Adverse Events of Special Interest (AESI)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Adverse events of special interest (AESIs) were collected.
Time Frame: Up to 153 weeks
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 4
Participants | 3

27. Secondary Outcome: CE Phase: Number of Participants With Adverse Events of Special Interest (AESI)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Adverse events of special interest (AESIs) were to be collected.
Time Frame: Up to 153 weeks
Population: No participants were enrolled in CE Phase as study was terminated.
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 0

28. Secondary Outcome: DE Phase: Number of Participants With Any Corneal Event by Maximum Grade as Per CTCAE Grade
Description: The corneal events were graded according to CTCAE version 5. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant. Higher grade indicates greater severity and an increase in CTCAE grade was defined relative to the Baseline grade. Results are presented for number of participants with any corneal events by maximum grade as per CTCAE grade.
Time Frame: Up to 153 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 4
Participants
  Grade 1 | 1
  Grade 2 | 0
  Grade 3 | 0

29. Secondary Outcome: CE Phase: Number of Participants With Any Corneal Events by Maximum Grade as Per CTCAE Grade
Description: The corneal events were to be graded according to CTCAE version 5. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant. Higher grade indicates greater severity and an increase in CTCAE grade was defined relative to the Baseline grade. Corneal Events were to be examined.
Time Frame: Up to 153 weeks
Population: No participants were enrolled in CE Phase as study was terminated.
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 0

30. Secondary Outcome: CE Phase: Progression-free Survival (PFS)
Description: PFS is defined as the time from randomization until the earliest date of confirmed progressive disease (PD) per IMWG, or death due to any cause.
Time Frame: Up to 153 weeks
Population: No participants were enrolled in CE Phase as study was terminated.
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 0

31. Secondary Outcome: CE Phase: Duration of Response (DoR)
Description: DoR is defined as the time from first documented evidence or PR or better until progressive disease per IMWG or death due to progressive disease among participants who achieve confirmed partial response or better.
Time Frame: Up to 153 weeks
Population: No participants were enrolled in CE Phase as study was terminated.
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 0

32. Secondary Outcome: CE Phase: Time to Response (TTR)
Description: TTR is defined as the time between the date of randomization and the first documented evidence of response (PR or better), among participants who achieve a response (confirmed PR or better).
Time Frame: Up to 153 weeks
Population: No participants were enrolled in CE Phase as study was terminated.
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 0

33. Secondary Outcome: CE Phase: Overall Survival (OS)
Description: OS is defined as the time from randomization until death due to any cause.
Time Frame: Up to 153 weeks
Population: No participants were enrolled in CE Phase as study was terminated.
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 0

34. Secondary Outcome: CE Phase: Number of Participants With AEs and SAEs
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that; results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations judged by physician, is associated with liver injury and impaired liver function. AEs and SAEs were to be coded using the Medical Dictionary for Regulatory Activities (MedDRA) coding system.
Time Frame: Up to 153 weeks
Population: No participants were enrolled in CE Phase as study was terminated.
Groups:
- 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab: Participants with Relapsed/Refractory Multiple Myeloma (RRMM) received 1.9 milligram (mg)/kilogram (kg) belantamab mafodotin intravenous (IV) infusion as powder for solution once every 3 weeks (Q3W) infused over 30- 60 minutes on day 1 of 21 day cycles in combination with 500 mg dostarlimab as a 30-minute IV infusion 1 hour after belantamab mafodotin end of infusion (EOI) on day 1 of 21 day cycles (Q3W).
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 0

35. Secondary Outcome: CE Phase: Number of Participants With AEs Leading to Discontinuation
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Number of participants with AEs leading to discontinuation were to be evaluated.
Time Frame: Up to 153 weeks
Population: No participants were enrolled in CE Phase as study was terminated.
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 0

36. Secondary Outcome: CE Phase: Number of Participants With Dose Reduction or Delay
Description: Number of participants with dose reduction or delay were to be evaluated.
Time Frame: Up to 153 weeks
Population: No participants were enrolled in CE Phase as study was terminated.
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 0

37. Secondary Outcome: CE Phase: Number of Participants With Clinically Significant Changes in Hematology Lab Parameters
Description: Blood samples were to be collected for the analysis of following hematology parameters: eosinophils, anemia, hemoglobin increased, lymphocyte count decreased, lymphocyte count increased, neutrophil count decreased, platelet count decreased, leukocytosis and white blood cell decreased. The laboratory parameters were to be graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5. Grade 1 (G1): mild; Grade 2 (G2): moderate; Grade 3 (G3): severe or medically significant. Higher grade indicates greater severity and an increase in CTCAE grade was defined relative to the Baseline grade.
Time Frame: Up to 153 weeks
Population: No participants were enrolled in CE Phase as study was terminated.
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 0

38. Secondary Outcome: CE Phase: Number of Participants With Clinically Significant Changes in Clinical Chemistry Lab Parameters
Description: Blood samples were to be collected for the analysis of following chemistry parameters: Hypoglycemia, hypoalbuminemia, alkaline phosphatase (ALP) increased, alanine aminotransferase (ALT) increased, aspartate aminotransferase (AST) increased, blood bilirubin increased, creatine kinase (CPK) increased, creatinine increased, gamma glutamyl transferase (GGT) increased, hyperkalemia, blood lactate dehydrogenase (LDH) increased, hypermagnesemia, hypomagnesemia, hypernatremia, hypercalcemia, hypocalcemia and chronic kidney disease. The laboratory parameters were to be graded according to CTCAE version 5. G1: mild; G2: moderate; G3: severe or medically significant. Higher grade indicates greater severity and an increase in CTCAE grade was defined relative to the Baseline grade.
Time Frame: Up to 153 weeks
Population: No participants were enrolled in CE Phase as study was terminated.
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All cause mortality, non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected maximum up to 153 weeks.
Description: Safety set included all participants who received at least 1 dose of any component of the combination therapy.
Arm/Group | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab
All-Cause Mortality (participants affected / at risk) | 2/4
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab (N=4)
Pyrexia (General disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1.9 mg/kg Belantamab Mafodotin + 500mg Dostarlimab (N=4)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Dry eye (Eye disorders) | 1 (2)
Eye irritation (Eye disorders) | 1 (2)
Foreign body sensation in eyes (Eye disorders) | 1 (2)
Vision blurred (Eye disorders) | 2 (7)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-01-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT06655818/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT06655818/SAP_001.pdf